CLINICAL TRIAL: NCT04300764
Title: Gamification to Increase Mobility in the Hospital
Acronym: Level Up
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was never launched due to COVID19 pandemic
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ryan Greysen, Ryan Greysen, MD, MHS, MA, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 834466
Record Dates: First submitted 2020-02-22; First posted 2020-03-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Coronary Heart Disease; Hypertension; Diabete Mellitus; Dyslipidemias; Obesity; Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Hypertension; Diabetes Mellitus; Dyslipidemias; Obesity; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will be recruited during an inpatient stay and given a Fitbit watch that will transmit data to the Way to Health study platform. Control participants' steps will be passively monitored. Data will continue to be collected for 30 days after discharge.
- Gamification Intervention (Experimental): Participants will be recruited during an inpatient stay and given a Fitbit watch that will transmit data to the Way to Health study platform. Intervention patients will receive daily text messages to help them set goals, receive feedback and support on their progress towards daily goals, and receive points for daily goals achieved. Data will continue to be collected for 30 days after discharge.
  Interventions: Behavioral: Gamification Intervention

INTERVENTIONS:
Behavioral: Gamification Intervention — Intervention participants will receive daily text messages to help them set goals, receive feedback and support on their progress towards daily goals, and receive points for daily goals achieved. Each participant will be given a Fitbit watch that will transmit data to the Way to Health study platform. Data will be passively collected during the inpatient stay and for 30 days after hospital discharge.
  Arms: Gamification Intervention

SUMMARY:
Low mobility is a mediator for poor outcomes of hospital care. Wearable devices will be used and 2-way texting via patient smartphones to monitor patients' physical activity during hospitalization with and without gamification to improve patient adherence to existing guidance on recommended activity. After discharge, investigators will assess patient care utilization (SNF, inpatient vs home rehab, ED visits, readmission) and conduct validated surveys on patient function at 30 days after discharge.

DETAILED DESCRIPTION:
Hospitalization is a common occurrence for older adults; approximately 6.8 million Medicare seniors experience an admission for acute care in any given year. This is often a sentinel event in the overall health trajectory of older adults that is complicated by functional impairment, Skilled Nursing Facility placement, and reduced mobility after discharge.

In the current paradigm, low mobility during hospitalization is largely viewed as a temporary inconvenience that should not affect overall functional ability or outcomes such nursing home placement and that patients should return to their previous activity level soon after they return home without lingering mobility changes. Recent research, however, suggests disruptions of basic activities of daily life such as mobility (getting out of bed and walking) may be "traumatic" or "toxic" to older adults with long-term post-hospital effects. What is lacked is precise data on how much immobility is noxious and how much mobility is needed to protect against adverse outcomes.

The primary objective is to assess the effectiveness of a gamification intervention to increase physical activity before hospital discharge. Investigators will explore patients' physical activity while in the hospital and if that differs across floors that have already deployed a nursing mobility protocol (Founders 10, 11, 12, 14). Investigators will also explore changes in patient functional status, SNF placement, and 30-day hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a medicine or cardiology floor in the hospital
* Age 50 years or older
* Have an AMPAC (mobility scale) score of greater than or equal to 21 or a Braden mobility sub-scale score of 4.

Exclusion Criteria:

* Inability to provide informed consent
* Does not have daily access to a smartphone compatible with the wearable device and not willing to use a device that the study team can provide
* Inpatient AMPAC score of less than 21 or a Braden mobility sub-scale score less than 4 indicating that independent physical activity may not be appropriate for the patient
* Are already enrolled in another physical activity study
* Any conditions that would prohibit participation in an inpatient physical activity program (at the discretion of attending physician or nurse caring for the patient in the hospital). To minimize the risk of contamination across study arms, we will only approach one patient per hospital room in shared rooms

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean daily step count during hospitalization | Average 5 days
  The primary outcome variable is the change in mean daily step count during hospitalization (from enrollment to discharge).

SECONDARY OUTCOMES:
Proportion of patients who attain pre-specified step thresholds during hospitalization and after discharge | Average 35 days
  Proportion of patients in each group who attain pre-specified step thresholds of 1000, 2000, 3000 during hospitalization and 3500, 4000, 4500, and 5000 after discharge
Hospital length of stay | Average 5 days
  Length of inpatient hospital stay
Discharge to post-acute facilities | 30 days
  Discharge to post-acute facilities (skilled nursing facility or rehabilitation facility)
30-day acute care utilization | 30 days
  30-day acute care utilization (hospital readmission or ED visits)
Change in activities of daily living | Average 35 days
  Change in functional status measure of activities of daily living from admission to 30 days post-discharge.using the Activities of Daily Living Scale.
Change in difficulty with walking | Average 35 days
  Change in functional status measure of difficulty with walking from admission to 30 days post-discharge using the Activities of Daily Living Scale.
Change in life space assessment | Average 35 days
  Change in functional status measure of life space assessment from admission to 30 days post-discharge.using the Life Space Activity Survey

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Greysen, MD, MHS, MA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States